CLINICAL TRIAL: NCT03063931
Title: Effect of the Oral Route of Magnesium on Pre and Post-mastectomy on the Post-surgery Pain
Brief Title: Pain and Magnesium
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHU-306; 2016-A01749-42 (Other: 2016-A01749-42)
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Neuropathic Pain Induced by Mastectomy
Keywords: Breast cancer; Mastectomy; Pain; Anxiety and Depression; Cognition; Quality of life
MeSH Terms: conditions — Breast Neoplasms; Pain; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- magnesium (Experimental)
  Interventions: Drug: Magnesium: Magnésium UPSA Action Continue®
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo: Lactose

INTERVENTIONS:
Drug: Magnesium: Magnésium UPSA Action Continue® — This clinical trial compares magnesium and placebo for the prevention of neuropathic pain induced by mastectomy assessed with a (0-10) numerical pain rating scale
  Arms: magnesium
Drug: Placebo: Lactose — This clinical trial compares magnesium and placebo for the prevention of neuropathic pain induced by mastectomy assessed with a (0-10) numerical pain rating scale
  Arms: placebo

SUMMARY:
In breast cancer patients undergoing a mastectomy, the aim of this study is to evaluate if the magnesium administered for 6 weeks starting two weeks before the surgery induces a decrease of pain intensity one month post-mastectomy compared to the placebo group.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled double-blind clinical trial conducted in the Oncology Hospital, Clermont-Ferrand, France, in 100 patients suffering from breast cancer and undergoing a total mastectomy.

This clinical trial compares magnesium and placebo for the prevention of neuropathic pain induced by mastectomy assessed with a (0-10) numerical pain rating scale. Cognition, anxiety, depression, sleep and quality of life are also assessed.

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥ 18 years,
* Patient with breast cancer who has a scheduled total mastectomy with or without treatment two weeks after inclusion with or without preoperative chemotherapy,
* Patient free from any new treatment or diet at the time of the inclusion,
* Cooperation and understanding sufficient to comply with the requirements of the study,
* Patients affiliated to the French Social Security,
* Patients with free and informed consent has been obtained

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients
* Patient with magnesemia >1,05 mmol/l
* Patient with severe renal insufficiency with creatinine clearance <30 ml min,
* Patient with an addiction to alcohol, as determined by the investigator,
* Diabetes (type I and II),
* Medical and surgical history incompatible with the study,
* Patient receiving treatment with Quinidine, L-Dopa,
* Childbearing age, no use of effective contraceptive method, pregnancy or lactation
* Patient exclusion period, or the total allowable compensation exceeded
* Patients undergoing a measure of legal protection (guardianship, supervision ...)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Measure of average pain intensity by a numerical rating scale | 5 days before the visit at 1 month post-mastectomy
  Measure of average pain intensity by a numerical rating scale assessed 5 days before the visit at 1 month post-mastectomy in magnesium and placebo groups.

SECONDARY OUTCOMES:
Pain assessment by the Neuropathic pain questionnaire | at month 1 and Month 3
Evaluation of analgesic consumption | at 3 month
Cognitive assessment by Trail Making Test A and B | at month 1 and month 3
Quality of life assessment by EORTC QLQ-C30 | at month 1 and month 3
Quality of life assessment by Pittsburg Sleep Quality Index (PSQI) | at month 1 and month 3
Anxiety and Depression assessment by DASS scale | at month 1 and month 3
Plasma and erythrocyte assays of magnesium | at inclusion visit, month 1 and month 3
Creatinine dosage | at inclusion visit
Urine assays of magnesium | at month 1 and month 3

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Morel V, Joly D, Villatte C, Pereira B, Pickering G. Preventive effect of oral magnesium in postmastectomy pain: protocol for a randomised, double-blind, controlled clinical trial. BMJ Open. 2018 Oct 4;8(9):e017986. doi: 10.1136/bmjopen-2017-017986. PMID 30287600